CLINICAL TRIAL: NCT00612430
Title: Phase II Trial of Bevacizumab Plus Etoposide for Patients With Recurrent Malignant Glioma
Brief Title: Ph II Bevacizumab + Etoposide for Pts w Recurrent MG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000379
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Results first posted 2013-07-26 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-05

CONDITIONS: Glioblastoma; Gliosarcoma
Keywords: Glioblastoma; Gliosarcoma; GBM; MG; Brain tumor; Bevacizumab; Avastin; Etoposide; VP-16; Etopophos; Toposar; VePesid; Glioblastoma multiforme; Recurrent GBM; Anaplastic astrocytoma; Malignant glioma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms; Astrocytoma; Glioma | interventions — Bevacizumab; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab + Etoposide (Experimental): Grade III and IV patients will receive: Bevacizumab administered intravenously at dose 10 mg/kg every two weeks. If patient tolerates 1st bevacizumab dose, subsequent doses may be given by local oncologists under direct supervision of Duke investigators. Etoposide administered orally, once daily for 1st 21 days of each 28-day treatment cycle. Dose of Etoposide will be 50 mg/m2/day.
  Interventions: Drug: Bevacizumab and Etoposide

INTERVENTIONS:
Drug: Bevacizumab and Etoposide — 32 pts w recurrent WHO grade III MG & 27 pts w recurrent WHO grade IV MG will be enrolled in this study. Estimated rate of accrual is 10 pts per month. The estimated date of study completion is 6-9 months from study initiation. Bevacizumab administered intravenously at dose 10 mg/kg every two weeks. If pt tolerates 1st bevacizumab dose, subsequent doses may be given by local oncologists under direct supervision of Duke investigators. Etoposide administered orally, once daily for 1st 21 days of each 28-day treatment cycle. Dose of Etoposide will be 50 mg/m2/day. The Duke investigators will review all la data & order treatment. Treatment will continue until either evidence of progressive disease, unacceptable toxicity, non-compliance w study follow-up, or withdrawal of consent.
  Other Names: Bevacizumab - Avastin; Etoposide-Etopophos-Toposar-VePesid-VP-16

SUMMARY:
Primary Objective to estimate 6-month progression free survival probability of patients with recurrent malignant glioma treated with Etoposide + Bevacizumab.

Secondary Objectives To evaluate safety & tolerability of Etoposide + Bevacizumab among patients with recurrent malignant glioma (RMG).

To evaluate radiographic response, progression free survival & overall survival of patients with recurrent malignant glioma treated with Etoposide + Bevacizumab.

DETAILED DESCRIPTION:
Exploratory, single-arm, ph II study designed to assess anti-tumor activity of combinatorial regimen consisting of Etoposide + Bevacizumab among patients with RMG. Primary endpoint of study is probability of progression-free survival at 6 months. Important secondary objective is to further assess safety of Etoposide & Bevacizumab for patients with recurrent malignant glioma.

If study demonstrates that combinatorial regimen of Etoposide + Bevacizumab is associated with encouraging anti-tumor activity among patients with RMG, further assessment of regimen in additional phase II & possibly phase III studies, will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Pts have confirmed diagnosis of recurrent/progressive WHO gr III & IV MG
* Age >18 rs
* Interval of >4 wks since prior surgery
* Interval of >4 wks since prior XRT/chemo, unless there is unequivocal evidence of progressive disease & pts have recovered from all anticipated toxicity of most recent therapy;
* Karnofsky performance status score >60
* Hematocrit >29 percent, ANC >1,500 cells/microliter, platelets >100,000 cells/microliter
* Serum creatinine <1.5 mg/dl, BUN <25 mg/dl, serum SGOT & bilirubin <1.5 x ULN
* For pts on corticosteroids, they have been on astable dose for 1wk prior to entry
* Signed informed consent approved by IRB prior to pt entry
* If sexually active, pts must agree to take contraceptive measures for duration of treatments.

Exclusion Criteria:

* Prior therapy w either bevacizumab/etoposide
* >3 prior recurrences
* Pregnancy/breast feeding
* Co-medication w immuno-suppressive agents other than corticosteroids including but not limited to cyclosporine, tacrolimus, sirolimus, mycophenolate mofetil
* Evidence of CNS hemorrhage on baseline MRI on CT scan
* Pts who require therapeutic anti-coagulation
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring IV antibiotics & psychiatric illness/social situations that would limit compliance w study requirements, or disorders associated w significant immunocompromised state
* Pts w another primary malignancy that has required treatment <past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-03; Primary Completion 2008-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Reardon, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- [Derived] Reardon DA, Desjardins A, Vredenburgh JJ, Gururangan S, Sampson JH, Sathornsumetee S, McLendon RE, Herndon JE 2nd, Marcello JE, Norfleet J, Friedman AH, Bigner DD, Friedman HS. Metronomic chemotherapy with daily, oral etoposide plus bevacizumab for recurrent malignant glioma: a phase II study. Br J Cancer. 2009 Dec 15;101(12):1986-94. doi: 10.1038/sj.bjc.6605412. Epub 2009 Nov 17. PMID 19920819
- See also: The Preston Robert Tisch Brain Tumor Center at DUKE — http://www.cancer.duke.edu/btc/

RESULTS

PARTICIPANT FLOW:
Groups:
- Grade III; Grade IV: Bevacizumab administered intravenously at dose 10 mg/kg every two weeks. If patient tolerates 1stbevacizumab dose, subsequent doses may be given by local oncologists under direct supervision of Duke investigators. Etoposide administered orally, once daily for 1st 21 days of each 28-day treatment cycle. Dose of Etoposide will be 50 mg/m2/day
Period: Overall Study
Arm/Group | Grade III | Grade IV
Started | 32 | 27
Completed | 32 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Grade III | Grade IV | Total
Number analyzed (Participants) | 32 | 27 | 59
Age Continuous [Median (Full Range); unit: years] | 45.9 (24.5-61.7) [24.5 to 61.7] | 54.3 (24.1-70.4) [24.1 to 70.4] | 48.5 (24.1-70.4) [24.1 to 70.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Progression-Free Survival (PFS)
Description: Percentage of participants surviving six months from the start of study treatment without progression of disease. PFS was defined as the time from the date of study treatment initiation to the date of the first documented progression. Progression was defined as greater than or equal to a 25% increase in the product of the largest perpendicular diameters of any enhancing lesion or any new enhancing tumor on MRI scans.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Grade III | Grade IV
Number analyzed (Participants) | 32 | 27
percentage of participants | 41 [24 to 57] | 44 [26 to 62]

2. Secondary Outcome: Objective Response Rate
Description: The percentage of participants with complete or partial response as determined by the following criteria: complete response was defined as complete disappearance on MR/CT of all enhancing tumor and mass effect, off all corticosteroids (or receiving only adrenal replacement doses), accompanied by a stable or improving neurologic examination; partial response was defined as greater than or equal to 50% reduction in tumor size on MR/CT by bi-dimensional measurement, on a stable or decreasing dose of corticosteroids, accompanied by a stable or improving neurologic examination. A confirmation of response was not required.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Grade III | Grade IV
Number analyzed (Participants) | 32 | 27
percentage of participants | 24 | 23

3. Secondary Outcome: Safety of Study Treatment Regimen
Description: Number of participants experiencing a non-hematologic toxicity ≥ grade 3 that was possibly, probably, or definitely related to study treatment.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Grade III | Grade IV
Number analyzed (Participants) | 32 | 27
participants | 9 | 13

4. Secondary Outcome: Median Progression-Free Survival
Description: Time in weeks from the start of study treatment to the date of first progression, or to death due to any cause. Patients alive who had not progressed as of the last follow-up had PFS censored at the last follow-up date. Median PFS was estimated using a Kaplan-Meier curve.
Time Frame: Patients were followed for a median of 91.4 weeks
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Grade III | Grade IV
Number analyzed (Participants) | 32 | 27
weeks | 24 [16 to 33] | 18 [13 to 40]

5. Secondary Outcome: Median Overall Survival (OS)
Description: Time in weeks from the start of study treatment to date of death due to any cause. Patients alive as of the last follow-up had OS censored at the last follow-up date. Median OS was estimated using a Kaplan-Meier curve.
Time Frame: median of 91.4 weeks
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Grade III | Grade IV
Number analyzed (Participants) | 32 | 27
weeks | 63.1 [36 to NA] — Follow-up was not long enough to provide an upper confidence limit for the median survival. | 46.4 [25 to 70]

ADVERSE EVENTS:
Time Frame: 2 years
Description: The adverse events were gathered in Common Terminology Criteria for Adverse Events v.3.0, and have been converted to v.4.0 for entry into ClinicalTrials.gov
Arm/Group | Grade III | Grade IV
Serious Adverse Events (participants affected / at risk) | 2/32 | 3/27
Other Adverse Events (participants affected / at risk) | 31/32 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Grade III (N=32) | Grade IV (N=27)
Colonic ulcer (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Stomach pain (Gastrointestinal disorders) | 1 | 0
Death NOS (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Grade III (N=32) | Grade IV (N=27)
Anemia (Blood and lymphatic system disorders) | 10 | 19
Cardiac disorders - Other, specify: S1-S2 with grade II/IV murmur (Cardiac disorders) | 0 | 1
Cardiac disorders - Other, specify: Variable Heart Rate (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, specify: Angina (Cardiac disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 2 | 0
Blurred vision (Eye disorders) | 5 | 3
Extraocular muscle paresis (Eye disorders) | 0 | 1
Eye disorders - Other, specify: Partial right homonymous hemianopsia (Eye disorders) | 1 | 0
Eye disorders - Other, specify: Visual acuity (Eye disorders) | 1 | 0
Eye disorders - Other, specify: Proptosis/enophthalmos (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 0 | 1
Flashing lights (Eye disorders) | 0 | 1
Night blindness (Eye disorders) | 0 | 1
Optic nerve disorder (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 1 | 0
Retinopathy (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 6 | 9
Diarrhea (Gastrointestinal disorders) | 7 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 3 | 0
Fecal incontinence (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 3 | 3
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 12 | 11
Nausea (Gastrointestinal disorders) | 11 | 6
Oral pain (Gastrointestinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 2
Rectal ulcer (Gastrointestinal disorders) | 1 | 1
Stomach pain (Gastrointestinal disorders) | 1 | 2
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 8 | 3
Edema face (General disorders) | 1 | 0
Edema limbs (General disorders) | 2 | 3
Fatigue (General disorders) | 17 | 17
Fever (General disorders) | 2 | 2
Gait disturbance (General disorders) | 4 | 3
Non-cardiac chest pain (General disorders) | 1 | 1
Pain (General disorders) | 1 | 2
Infections and infestations - Other, specify: Lung Abcess (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify: Bronchitis (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 3 | 2
Nail infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 3 | 1
Skin infection (Infections and infestations) | 0 | 3
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 6 | 8
Alkaline phosphatase increased (Investigations) | 0 | 5
Aspartate aminotransferase increased (Investigations) | 3 | 3
Blood bilirubin increased (Investigations) | 0 | 3
Cholesterol high (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 17 | 18
Platelet count decreased (Investigations) | 6 | 14
Weight gain (Investigations) | 2 | 0
Weight loss (Investigations) | 3 | 2
White blood cell decreased (Investigations) | 17 | 22
Anorexia (Metabolism and nutrition disorders) | 6 | 7
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 9 | 17
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 2
Hypernatremia (Metabolism and nutrition disorders) | 0 | 4
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 7
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 6
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 6
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 3 | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 | 5
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Ataxia (Nervous system disorders) | 8 | 13
Cognitive disturbance (Nervous system disorders) | 12 | 12
Depressed level of consciousness (Nervous system disorders) | 11 | 9
Dizziness (Nervous system disorders) | 5 | 4
Dysgeusia (Nervous system disorders) | 1 | 0
Dysphasia (Nervous system disorders) | 7 | 9
Encephalopathy (Nervous system disorders) | 0 | 1
Facial nerve disorder (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 13 | 9
Intracranial hemorrhage (Nervous system disorders) | 3 | 0
Memory impairment (Nervous system disorders) | 6 | 13
Nervous system disorders - Other, specify: Mood alteration, NOS (Nervous system disorders) | 0 | 2
Nervous system disorders - Other, specify: Fell; hematoma on scalp (Nervous system disorders) | 1 | 0
Nervous system disorders - Other, specify: Peripheral neuropathy (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Oculomotor nerve disorder (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 6 | 12
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 8
Seizure (Nervous system disorders) | 8 | 4
Tremor (Nervous system disorders) | 1 | 9
Agitation (Psychiatric disorders) | 0 | 4
Anxiety (Psychiatric disorders) | 4 | 1
Confusion (Psychiatric disorders) | 3 | 9
Depression (Psychiatric disorders) | 0 | 4
Insomnia (Psychiatric disorders) | 8 | 8
Psychosis (Psychiatric disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 11 | 3
Urinary frequency (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 4
Urinary retention (Renal and urinary disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 1
Reproductive system and breast disorders - Other, specify: Sexual Dysfunction, NOS (Reproductive system and breast disorders) | 6 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 2
Skin and subcutaneous tissue disorders - Other, specify: Folliculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify: Sore behind ear (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify: Petechiae/purpura- face all over (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flashes (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 10 | 7
Hypotension (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No